CLINICAL TRIAL: NCT06081101
Title: Ultrasound Guided Sacroiliac Joint Injections With Ketorolac Versus Corticosteroid: A Prospective Non-inferiority Study
Brief Title: Ketorolac Versus Corticosteroid Injections for Sacroiliac Joint Pain
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: McMaster_University_KVC
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sacro-iliac Joint Pain
MeSH Terms: interventions — Methylprednisolone; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Corticosteroid (Active Comparator): Patients will receive ultrasound guided corticosteroid injection to see pain relief after injection
  Interventions: Drug: Methylprednisolone Injection
- Ketorolac (Active Comparator): Patients will receive ultrasound guided ketorolac injection to see pain relief after injection
  Interventions: Drug: Ketorolac Injection

INTERVENTIONS:
Drug: Methylprednisolone Injection — Medication will be injected into SI joint under ultrasound guidance
  Arms: Corticosteroid
Drug: Ketorolac Injection — Medication will be injected into SI joint under ultrasound guidance
  Arms: Ketorolac

SUMMARY:
This study will contribute to the current literature that have compared joint injections with steroid versus ketorolac providing evidence for the use of ketorolac for SI joint pain. Currently steroid is the clinical standard for joint injections, however with repetitive use, steroid injections can damage the joint. Ketorolac is an alternative anti-inflammatory medication that does not cause the same joint damage and at a cheaper cost than steroid. The investigators hypothesize that ultrasound guided SI joint injections utilizing ketorolac provide the same pain relief as corticosteroid SI joint injections measured at 2, 6 and 12 weeks post injection. This would allow more frequent injections to control pain at a decreased cost to the healthcare system.

DETAILED DESCRIPTION:
The majority of people will suffer from low back pain at some point in their life with 15-25% of axial low back pain originating at the sacroiliac (SI) joint. This pain is thought to be due to inflammation of the SI joint capsule, ligaments or bone. Following conservative management strategies such as mobility work, core strengthening and physiotherapy, as well as pharmacologic management, an SI joint injection would be the next treatment modality. Corticosteroid injections are currently the standard of care for joint injections. The corticosteroid minimizes pain by interrupting the bodies inflammatory cascade primarily by inhibiting the phospholipase A2 enzyme. However, with repetitive use, steroids can cause cartilaginous damage of the joint. With chondrocyte dysfunction being a key part of early osteoarthritis, these injections may expedite the arthritic joint changes. Due to this damage, physicians try to spread out joint injections as far as possible to reduce this risk even if the patient begins to experience more severe joint pain.

One possible alternative to steroids is the use of ketorolac, an non-steroidal anti-inflammatory drug (NSAID). Ketorolac joint injections have been shown to have similar pain reducing effects to steroids when used for shoulder, knee, hip and carpometacarpal joint pain. They have also been used widely in the National Football League to treat musculoskeletal injuries and in the post-operative phase to reduce opioid usage to manage pain. NSAIDS provide analgesia by inhibiting the cyclooxygenase (COX) family of enzymes that are involved with formation of prostaglandins. These prostaglandins are inflammatory mediators that promote inflammation and activates nociceptive neurotransmitters. Although there are known side effects of NSAIDs including increasing propensity for GI bleeds, kidney and liver disease, joint injections may have less systemic side effects compared to their oral counterparts. Another benefit of Ketorolac is the fact it is significantly cheaper than steroids. With less chondrotoxic effects, perhaps Ketorolac injections could be administered more frequently, not allowing the patient to have increasing pain levels, at less cost to the health care system even with more frequent administration.

ELIGIBILITY:
Inclusion Criteria:

* SI joint pain for at least 3 months
* Age greater than 18
* Must have at least 3 special tests positive for SI joint pain on physical exam

Exclusion Criteria:

* Previous back surgery
* Radicular leg pain
* Discogenic pain
* Myofascial pain syndrome
* Depression
* Systemic infection or localized infection at anticipated needle entry sites
* Cognitive impairment preventing informed consent or accurate collection of data
* Patient allergic to medication used
* NSAID contraindications including:
* Gastrointestinal bleeds
* Renal failure
* Symptomatic congestive heart failure
* Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sacroiliac (SI) joint pain | 3 months following SI joint injection
  SI joint pain at 2, 6 and 12 week marks post SI joint injection measured on visual analogue scale. Higher numbers equate to worse pain and worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael G. DeGroote Pain Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participant data will be kept on an encrypted device. Patient identifiers will not be used as patient will be matched with a randomized patient ID

REFERENCES:
- [Background] Park KD, Kim TK, Bae BW, Ahn J, Lee WY, Park Y. Ultrasound guided intra-articular ketorolac versus corticosteroid injection in osteoarthritis of the hip: a retrospective comparative study. Skeletal Radiol. 2015 Sep;44(9):1333-40. doi: 10.1007/s00256-015-2174-9. Epub 2015 Jun 3. PMID 26031217
- [Background] Aranke M, McCrudy G, Rooney K, Patel K, Lee CA, Hasoon J, Kaye AD. Minimally Invasive and Conservative Interventions for the Treatment of Sacroiliac Joint Pain: A Review of Recent Literature. Orthop Rev (Pavia). 2022 May 31;14(4):34098. doi: 10.52965/001c.34098. eCollection 2022. PMID 35769646
- [Background] Koh SH, Lee SC, Lee WY, Kim J, Park Y. Ultrasound-guided intra-articular injection of hyaluronic acid and ketorolac for osteoarthritis of the carpometacarpal joint of the thumb: A retrospective comparative study. Medicine (Baltimore). 2019 May;98(19):e15506. doi: 10.1097/MD.0000000000015506. PMID 31083191
- [Background] Shapiro PS, Rohde RS, Froimson MI, Lash RH, Postak P, Greenwald AS. The effect of local corticosteroid or ketorolac exposure on histologic and biomechanical properties of rabbit tendon and cartilage. Hand (N Y). 2007 Dec;2(4):165-72. doi: 10.1007/s11552-007-9042-6. Epub 2007 May 5. PMID 18780047
- [Background] Beitzel K, McCarthy MB, Cote MP, Apostolakos J, Russell RP, Bradley J, ElAttrache NS, Romeo AA, Arciero RA, Mazzocca AD. The effect of ketorolac tromethamine, methylprednisolone, and platelet-rich plasma on human chondrocyte and tenocyte viability. Arthroscopy. 2013 Jul;29(7):1164-74. doi: 10.1016/j.arthro.2013.04.006. PMID 23809450
- [Background] Cooke C, Osborne J, Jackson N, Keating P, Flynn J, Markel D, Chen C, Lemos S. Acetaminophen, bupivacaine, Duramorph, and Toradol: A comparison of chondrocyte viability and gene expression changes in osteoarthritic human chondrocytes. Knee. 2020 Dec;27(6):1746-1752. doi: 10.1016/j.knee.2020.10.019. Epub 2020 Nov 13. PMID 33197813
- [Background] Xu J, Qu Y, Li H, Jiang T, Zheng C, Wang B, Shen P. Effect of ketorolac in intra-articular injection analgesia for postoperative pain in patients undergoing shoulder arthroscopy: a pilot-controlled clinical study. J Pain Res. 2019 Jan 17;12:417-422. doi: 10.2147/JPR.S178413. eCollection 2019. PMID 30705607
- [Background] Taheri P, Dehghan F, Mousavi S, Solouki R. Comparison of Subacromial Ketorolac Injection versus Corticosteroid Injection in the Treatment of Shoulder Impingement Syndrome. J Res Pharm Pract. 2017 Oct-Dec;6(4):223-227. doi: 10.4103/jrpp.JRPP_17_57. PMID 29417082
- [Background] Matava M, Brater DC, Gritter N, Heyer R, Rollins D, Schlegel T, Toto R, Yates A. Recommendations of the national football league physician society task force on the use of toradol((R)) ketorolac in the national football league. Sports Health. 2012 Sep;4(5):377-83. doi: 10.1177/1941738112457154. PMID 23016110
- [Background] Barkho JO, Li YK, Duku E, Thoma A. Ketorolac May Increase Hematoma Risk in Reduction Mammaplasty: A Case-control Study. Plast Reconstr Surg Glob Open. 2018 Mar 19;6(3):e1699. doi: 10.1097/GOX.0000000000001699. eCollection 2018 Mar. PMID 29707458
- [Background] Jurgensmeier K, Jurgensmeier D, Kunz DE, Fuerst PG, Warth LC, Daines SB. Intra-articular Injections of the Hip and Knee With Triamcinolone vs Ketorolac: A Randomized Controlled Trial. J Arthroplasty. 2021 Feb;36(2):416-422. doi: 10.1016/j.arth.2020.08.036. Epub 2020 Aug 22. PMID 32950343
- [Background] Piuzzi NS, Ng M, Kantor A, Ng K, Kha S, Mont MA, Muschler GF. What Is the Price and Claimed Efficacy of Platelet-Rich Plasma Injections for the Treatment of Knee Osteoarthritis in the United States? J Knee Surg. 2019 Sep;32(9):879-885. doi: 10.1055/s-0038-1669953. Epub 2018 Sep 6. PMID 30189436
- [Background] Bellamy JL, Goff BJ, Sayeed SA. Economic Impact of Ketorolac vs Corticosteroid Intra-Articular Knee Injections for Osteoarthritis: A Randomized, Double-Blind, Prospective Study. J Arthroplasty. 2016 Sep;31(9 Suppl):293-7. doi: 10.1016/j.arth.2016.05.015. Epub 2016 May 18. PMID 27402605
- [Background] D'Arcy Y, Mantyh P, Yaksh T, Donevan S, Hall J, Sadrarhami M, Viktrup L. Treating osteoarthritis pain: mechanisms of action of acetaminophen, nonsteroidal anti-inflammatory drugs, opioids, and nerve growth factor antibodies. Postgrad Med. 2021 Nov;133(8):879-894. doi: 10.1080/00325481.2021.1949199. Epub 2021 Jul 12. PMID 34252357
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210